CLINICAL TRIAL: NCT02264028
Title: Metabolism and Pharmacokinetics of [14C]-DK-AH 269 CL After Administration of Single Doses of 5 mg [14C]-DK-AH 269 CL Intravenously and 10 mg [14C]-DK-AH 269 CL as Oral Solution in a Parallel-group Design in 12 Healthy Male Volunteers
Brief Title: Metabolism and Pharmacokinetics of [14C]-DK-AH 269 CL in 12 Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 503.209
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions

ARMS (2):
- [14C]-DK-AH 269 CL intravenous (Active Comparator)
  Interventions: Drug: [14C]-DK-AH 269 CL, solution for infusion
- [14C]-DK-AH 269 CL oral (Experimental)
  Interventions: Drug: [14C]-DK-AH 269 CL, drinking solution

INTERVENTIONS:
Drug: [14C]-DK-AH 269 CL, solution for infusion
  Arms: [14C]-DK-AH 269 CL intravenous
Drug: [14C]-DK-AH 269 CL, drinking solution
  Arms: [14C]-DK-AH 269 CL oral

SUMMARY:
* To investigate absorption, metabolism and excretion of [14C]-DK-AH 269 CL after oral and intravenous administration in healthy volunteers
* To assess the safety and tolerability of DK-AH 269 CL after oral and intravenous administration to healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* 50 to 65 years of age
* Body Mass Index (BMI) of 19.9 to 29.9 kg/m2
* Resting heart rate (HR) (after 5 min. in the supine position) of more than 55 bpm
* All volunteers will have given their written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion Criteria:

* Any finding at the medical examination (including BP, HR and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, hematological/oncological, immunological or hormonal disorders
* Diseases of the central nervous system or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial within two weeks prior to administration or during the trial
* Participation in another trial with an investigational drug (≤ two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within 2 months prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range and of clinical relevance
* Inability to comply with dietary regimen of study centre

Not necessarily clinically relevant abnormalities, but specific exclusion criteria for the drugs under study or for the study:

* Subjects at increased risk for development of cardiac arrhythmia (e.g. family history of long QT syndrome or sudden cardiac death)
* ECG: PR interval > 210 ms
* HR at rest ≤ 55 beats per minute (bpm)
* Relevant ophthalmological disease

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-03; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of the analytes in plasma (Cmax) | Up to 96 hours after start of treatment
Area under the concentration-time curve of the analytes in plasma (AUC) | Up to 96 hours after start of treatment
Time from dosing to the maximum concentration of the analytes in plasma (tmax) | Up to 96 hours after start of treatment
Terminal rate constant of the analytes in plasma (λz) | Up to 96 hours after start of treatment
Terminal half-life of the analytes in plasma (t1/2) | Up to 96 hours after start of treatment
Mean residence time of the analytes in the body after intravenous administration (MRT) | Up to 96 hours after start of treatment
Mean residence time of the analytes in the body after oral administration (MRTpo) | Up to 96 hours after start of treatment
Apparent clearance of the analytes in plasma following extravascular administration (CL/F) | Up to 96 hours after start of treatment
Total clearance of the analytes in plasma following intravascular administration (CL) | Up to 96 hours after start of treatment
Apparent volume of distribution of the analytes during the terminal phase λz following extravascular administration (Vz/F) | Up to 96 hours after start of treatment
Volume of distribution at steady state (Vss) | Up to 96 hours after start of treatment
Fraction of analytes eliminated in urine from 0 to the time of the last quantifiable data point (fe0-tz) | Up to 120 hours after start of treatment
Fraction of analytes eliminated in faeces from 0 to the time of the last quantifiable data point (fefaeces,0-tz) | Up to 120 hours after start of treatment
Renal clearance of the analytes from 0 to the time of the last quantifiable data point (CLR,0-tz) | Up to 120 hours after start of treatment
Fraction of dose absorbed, based on radioactivity data (Fa) | Up to 96 hours after start of treatment
Absolute bioavailability of the analytes after oral administration (F) | Up to 96 hours after start of treatment
Ratio of CBlood cells/Cplasma [14C]-radioactivity | Up to 96 hours after start of treatment
Number of patients with clinically significant findings in vital signs | up to 12 days after last drug administration
  blood pressure, heart rate
Number of patients with clinically significant findings in 12-lead ECG | up to 12 days after last drug administration
Number of patients with clinically significant findings in 2-lead ECG (telemetry) | up to 90 minutes after start of treatment
Clinically significant changes from baseline in physical examination | Pre-dose, and 12 days after last drug administration
Occurrence of visual phenomena | up to 120 hours after start of treatment
  questionnaire
Number of patients with clinically significant findings in clinical laboratory tests | up to 12 days after last drug administration